CLINICAL TRIAL: NCT02351063
Title: HF Assessment With BNP in the Home: Part II
Acronym: HABIT-II
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor's discretion to terminate study prematurely for further evaluation.
Sponsor: Alere San Diego (Industry)
Responsible Party: Sponsor
Organization: Abbott RDx Cardiometabolic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BSTE-0144
Record Dates: First submitted 2015-01-12; First posted 2015-01-30 (Estimated); Results first posted 2019-02-04 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Heart Failure
Keywords: Heart failure; BNP; home testing; remote monitoring
MeSH Terms: conditions — Heart Failure | interventions — Diuretics; Adrenergic beta-Antagonists; Angiotensin-Converting Enzyme Inhibitors; Angiotensin Receptor Antagonists; Mineralocorticoid Receptor Antagonists; Vasodilator Agents; Nitrates

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Daily BNP (Experimental): Subjects will be asked to test their BNP at home every day for a period of 180 days using the AlereTM HeartCheck System (the Test System). In addition to BNP, weights and signs and symptoms of HF will be collected each day of testing. The HeartCheck data is transmitted via a secure wireless protocol to the HealthCOM health monitoring portal where it is available to the medical staff. The subject's's physician and medical staff will be required to evaluate the data and determine if a change in HF treatment is advisable. All changes of heart failure medications are at the discretion of the treating physician and medical staff of the institution.
  Interventions: Drug: Changes of heart failure medications

INTERVENTIONS:
Drug: Changes of heart failure medications — Changes in dosage of existing medications or introduction of new medications to improve heart failure condition.
  Other Names: Diuretics; Beta blockers; ACE inhibitors; Angiotensin II receptor antagonists; Aldosterone antagonists; Vasodilators; Nitrates; Inotropes; Other HF mediations

SUMMARY:
HABIT-II is a feasibility study aimed at home monitoring of patients with heart failure. B-type natriuretic peptide (BNP) has strong correlations to the severity of heart failure. Lower BNP levels are closely associated with better clinical outcomes. The goal of HABIT-II is to demonstrate that the results of daily patient self-testing of BNP at home will provide sufficient information to guide physicians to modify therapy and lower BNP levels over time.

DETAILED DESCRIPTION:
This is a single arm multi-center pilot study. Subjects with heart failure (HF) who are discharged following an acute decompensated heart failure (ADHF) event and subjects who are seen as outpatients with worsening signs or symptoms of HF, who meet enrollment criteria, are candidates for this study. Subjects with HF with reduced left ventricular ejection fraction (HFREF) and subjects with HF with preserved ejection fraction (HFPEF) are eligible. The eventual objective of this area of research is to demonstrate that HF subjects assisted by frequent B-type natriuretic peptide (BNP) measurements integrated into a home health management system have improved clinical outcomes. The specific objective of this study is to demonstrate that frequent BNP measurements integrated into a home health management system used by physicians to modify or intensify therapy will lead to a reduced risk of ADHF events as measured by a reduction in BNP levels. Subjects will be asked to test their BNP at home every day for a period of 180 days using the AlereTM HeartCheck System (the Test System). In addition to BNP, weights and signs and symptoms of HF will be collected each day of testing. The HeartCheck data is transmitted via a secure wireless protocol to the HealthCOM health monitoring portal where it is available to the medical staff.

Enrollment goal is 110 evaluable subjects. Potential subjects who meet the study's inclusion and exclusion criteria will be interviewed about their interest in participating in the study. Potential subjects that show interest in the study will be judged for their willingness, ability and reliability to perform fingerstick BNP measurements every day for 180 days while at home and be able to report the results using the HeartCheck system. All qualifying subjects who agree to participate and provide Informed Consent will be trained to use the HeartCheck system which includes daily BNP measurements, daily body weight measurements, and daily health survey questions. Subjects who successfully complete their training will be judged on their proficiency in all study activities. If found to be proficient; they will use the system at home. After a short lead-in period, an algorithm (similar in concept to a moving average) will be applied to the BNP data resulting in a BNP-based parameter and alerts will be created when this parameter is rising, or during periods of sustained high BNP. The patient's physician and medical staff will be required to evaluate all BNP based alert notifications and determine if a change in HF treatment is advisable. All changes in HF treatment, with or without BNP-based alerts, are at the discretion of the treating physician and medical staff of the institution.

The primary endpoint of the study is a significant lowering of BNP across the population. At approximately 1, 3 and 6 months after enrollment, subjects will return to the clinic for physical examination, clinical assessment, and review of interval medical status by their health care provider. In addition, if warranted, a home health care professional may visit the subject at home at any time during the study when additional counseling or training may be of benefit for compliance to the protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Adults at least 18 years of age
2. Willing to sign an Informed Consent Form
3. Ambulatory subjects with worsening HF defined as:

   1. Admitted to the hospital or treated in an outpatient clinic with a diagnosis of decompensated HF for which treatment will be administered; or
   2. Seen in an outpatient setting (i.e. heart failure clinic, general practice or cardiology office, urgent care unit) with a documented history of HF and with signs of worsening HF condition or decompensation, where worsening HF condition is defined as one or more of the following;

   i. Increase in NYHA class with worsening symptoms (i.e. dyspnea, fatigue) at same level of activity

   ii. Symptoms requiring change in dosage of one or more HF medication.

   iii. - Physical evaluation consistent with worsening HF signs (i.e. elevated jugular vein pressure (JVP), ankle edema, dyspnea, abdominal distension, >4 lb. or >1.8 kg weight increase in past week)
4. Must have some documented evidence of their current LVEF status as < 40% or > 40% (preferably a determination of %LVEF) at the time they begin BNP self-testing or within 2 months of enrollment
5. At least one BNP value during the index hospitalization or within 2 weeks of the index visit to clinic with worsening HF that meet the following criteria

   1. 400 pg/mL BNP (3200 pg/mL NT-proBNP) for subjects diagnosed with HFREF (LVSD < 40%) adjusted for BMI > 35
   2. 300 pg/mL BNP (2400 pg/mL NT-proBNP) for subjects diagnosed with HFPEF (LVSD > 40%) adjusted for BMI > 35
6. Deemed willing and suitable for HeartCheck BNP home testing and participation in this study;

   AND
7. Successfully trained and deemed proficient on how to perform a fingerstick and to use the HeartCheck system.

Exclusion Criteria:

1. Primary diagnosis at presentation of the index event of Acute Coronary Syndrome (ACS) (myocardial infarction (MI) or unstable angina).
2. Prior heart transplant or planned transplant within the next 3 months
3. Current or planned use of left ventricular assist device (LVAD) within 3 months
4. Current or planned inotrope dependent therapy within 3 months
5. Current or planned percutaneous coronary intervention (PCI) or coronary artery bypass graft (CABG) within 3 months
6. Life expectancy less than 6 months for causes other than for cardiovascular reasons
7. End stage renal disease (estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m2)
8. Other misc. cardiovascular and non-cardiovascular conditions such as amyloidosis, infiltrative cardiomyopathy, peripartum cardiomyopathy unless present for at least 12 months, acute myocarditis
9. Receiving investigational medications or therapy
10. Hematocrit known to be outside the 25-50% range of the HeartCheck system requirements
11. Deemed likely to be noncompliant with protocol by the Investigator
12. Residence in regions where transmission of test data or home visits are not possible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2014-04; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Maisel, MD, Principal Investigator — San Diego Veterans Administration Medical Center; Ken McDonald, MD, Principal Investigator — St Vincent's University Hospital, Ireland
Locations (13):
- United States (6):
  - Veterans Administration Medical Center, Loma Linda, California
  - Veterans Administration Medical Center, San Diego, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Veterans Administration Medical Center, Minneapolis, Minnesota
  - Ohio State University Medical Center, Columbus, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
- St. Michael's Hospital, Dublin, Dun Laoghaire, Ireland
- University Medical Center Groningen, Groningen, Netherlands
- New Zealand (2):
  - University of Auckland, Auckland
  - Christchurch Hospital, Christchurch
- Universitetssjukhuset Linköping, Linköping, Sweden
- United Kingdom (2):
  - Western Infirmary, Glasgow
  - Kings College, London

REFERENCES:
- [Background] Maisel A, Barnard D, Jaski B, Frivold G, Marais J, Azer M, Miyamoto MI, Lombardo D, Kelsay D, Borden K, Iqbal N, Taub PR, Kupfer K, Clopton P, Greenberg B. Primary results of the HABIT Trial (heart failure assessment with BNP in the home). J Am Coll Cardiol. 2013 Apr 23;61(16):1726-35. doi: 10.1016/j.jacc.2013.01.052. Epub 2013 Mar 26. PMID 23500322
- [Background] Januzzi JL Jr, Rehman SU, Mohammed AA, Bhardwaj A, Barajas L, Barajas J, Kim HN, Baggish AL, Weiner RB, Chen-Tournoux A, Marshall JE, Moore SA, Carlson WD, Lewis GD, Shin J, Sullivan D, Parks K, Wang TJ, Gregory SA, Uthamalingam S, Semigran MJ. Use of amino-terminal pro-B-type natriuretic peptide to guide outpatient therapy of patients with chronic left ventricular systolic dysfunction. J Am Coll Cardiol. 2011 Oct 25;58(18):1881-9. doi: 10.1016/j.jacc.2011.03.072. PMID 22018299
- [Background] Motiwala SR, Januzzi JL Jr. Using biomarkers to "guide" heart failure management: current perspectives and future directions. Cardiol Rev. 2013 May-Jun;21(3):127-34. doi: 10.1097/CRD.0b013e3182769073. PMID 23032578
- [Background] Maisel A, Mueller C, Adams K Jr, Anker SD, Aspromonte N, Cleland JG, Cohen-Solal A, Dahlstrom U, DeMaria A, Di Somma S, Filippatos GS, Fonarow GC, Jourdain P, Komajda M, Liu PP, McDonagh T, McDonald K, Mebazaa A, Nieminen MS, Peacock WF, Tubaro M, Valle R, Vanderhyden M, Yancy CW, Zannad F, Braunwald E. State of the art: using natriuretic peptide levels in clinical practice. Eur J Heart Fail. 2008 Sep;10(9):824-39. doi: 10.1016/j.ejheart.2008.07.014. Epub 2008 Aug 29. PMID 18760965
- [Background] Troughton RW, Frampton CM, Yandle TG, Espiner EA, Nicholls MG, Richards AM. Treatment of heart failure guided by plasma aminoterminal brain natriuretic peptide (N-BNP) concentrations. Lancet. 2000 Apr 1;355(9210):1126-30. doi: 10.1016/s0140-6736(00)02060-2. PMID 10791374

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Daily BNP
Started | 1
Completed | 1 (Study terminated. No study data collected.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: One subject enrolled but no data collected. Study terminated by sponsor.
Arm/Group | Daily BNP
Number analyzed (Participants) | 0
Age, Categorical
Sex: Female, Male
Race and Ethnicity Not Collected — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change in BNP
Description: After a short lead-in period, an algorithm (similar in concept to a moving average) will be applied to the BNP data resulting in a BNP-based parameter. The primary endpoint of the study is a significant lowering of BNP across the population, such that values for the population are reduced to levels below a predetermined threshold and kept below the threshold for the duration of subsequent testing and observation.
Time Frame: 6 months
Population: One subject enrolled but no data collected. Study terminated by sponsor.
Groups:
- All Subjects: One subject enrolled but no data collected. Study terminated by sponsor.
Arm/Group | All Subjects
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | All Subjects
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No